CLINICAL TRIAL: NCT01064583
Title: Long-term Effect of Dietary Intervention With Flavanol-containing Cocoa on Vascular Function of Diabetic Patients
Brief Title: Cocoa Flavanols and Painfree Walking Distance
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Klinik für Kardiologie, Pneumologie und Angiologie, Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Flavanols-PAD
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Peripheral Artery Disease; Diabetes Mellitus
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus | interventions — Chocolate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- flavanol rich cocoa drink (596mg) (Experimental): dissolved in water, twice daily intervention
  Interventions: Other: cocoa
- flavanol poor cocoa drink ( 13mg) (Experimental): dissolved in water, twice daily intervention
  Interventions: Other: cocoa

INTERVENTIONS:
Other: cocoa — dissolved in water twice-daily intervention

SUMMARY:
To characterize potential vascular long-term effects of flavanols in patients with peripheral artery occlusive disease (PAOD), a placebo-controlled double-blinded randomized control study will be performed in 62 patients randomized in two groups. Patients will twice daily receive either a flavanol-poor cocoa drink or a flavanol-rich cocoa drink over a period of 60 days months.

DETAILED DESCRIPTION:
62 Type 2 diabetics according to the criteria of the American Diabetes Association suffering from PAOD with a pain free walking distance less than 250m will be enrolled.

Patients will twice daily receive either a flavanol-poor cocoa drink (13mg/dl)or a flavanol-rich cocoa drink (596mg/dl) over a period of 60 days.

The general condition, the pain free walking distance and the vascular function measured by Doppler Ultrasound will be determined before and two month after cocoa ingestion

ELIGIBILITY:
Inclusion Criteria:

* peripheral artery disease (Fontaine IIb)
* diabetes mellitus
* > 18 years

Exclusion Criteria:

* acute and terminal renal failure
* acute infection
* heart failure (NYHA III-IV)
* arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-10; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
painfree walking distance | 60 days

SECONDARY OUTCOMES:
endothelial function | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Christian Heiss, MD, Principal Investigator — Heinrich Heine University; Malte Kelm, MD, Study Chair — Heinrich Heine University
Locations (1):
- Heinrich Heine University, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- See also: Related Info — http://www.uniklinik-duesseldorf.de/kardiologie